CLINICAL TRIAL: NCT05450523
Title: Neutrophil Gelatinase-Associated Lipocalin (NGAL) Rapid Test (Colloidal Gold)
Brief Title: Neutrophil Gelatinase-Associated Lipocalin (NGAL) Rapid Test (Colloidal Gold) Clinical Trial Protocol
Status: Completed | Type: Observational
Sponsor: Qingdao HIGHTOP Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HT1.0
Record Dates: First submitted 2022-06-27; First posted 2022-07-08 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Peritoneal Dialysis-associated Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the requirements of the "Technical Guidelines for Clinical Trials of In Vitro Diagnostic Reagents", the first registered product (hereinafter referred to as the assessment reagent) - Neutrophil Gelatinase-Associated Lipocalin (NGAL) Rapid Test (Colloidal Gold) was tested in clinical institutions. ) for clinical validation trials. Prove that the clinical performance of the assessment reagent meets the requirements of the intended use.

ELIGIBILITY:
Inclusion Criteria:

Patients treated with peritoneal dialysis due to kidney disease, including those with confirmed peritonitis and those without peritonitis. There are no age or gender requirements, and informed consent is required.

Exclusion Criteria:

1. Patients who have been treated with antibiotics for peritonitis before taking the sample.
2. Incomplete information, including: sample ID number, gender, age, department, clinical diagnosis, sample type, and sampling date.
3. The sample size is insufficient.
4. Repeated cases.
5. The samples whose permeate is red in visual inspection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with peritoneal dialysis due to kidney disease, including those with confirmed peritonitis and those without peritonitis.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Assessment reagent test results and clinical reference standard statistics | 8 months
  The peritoneal dialysis effluent collected from the subjects was tested blindly with the assessment reagents, and the test results were compared with the clinical reference standards. By evaluating the clinical sensitivity and specificity of the assessment reagents, the feasibility of clinical application of the assessment reagents was evaluated.
Statistical analysis of non-professional self-testing test | 8 months
  There is no need to train non-professionals. After reading the instructions and labels, non-professionals can evaluate their ability to understand key information such as instructions and packaging labels through questionnaires; Research, comparison of test results of different forms of reagents, and comparison with professional test results to evaluate their operational capabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Qinkai Chen, Chief physician, Study Chair — The first affiliated hosital of Nangchang university
Locations (1):
- The first affiliated hosital of Nangchang university, Nanchang, Jiangxi, China